CLINICAL TRIAL: NCT04429425
Title: A Prospective Randomized Comparative Study of Effectiveness of Epidural Anesthesia to Reduce Postoperative Ileus in Patients Undergoing Colorectal Surgery.
Brief Title: Does Epidural Anesthesia Reduce Postoperative Ileus Following Colorectal Surgery?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pinar Yazici, Assoc Prof, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-EPI-CRS-2020
Record Dates: First submitted 2020-03-17; First posted 2020-06-12 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Disorders; Postoperative Ileus
Keywords: colorectal surgery; postoperative ileus; epidural anesthesia; enhanced recovery after surgery
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: each patient will be randomly asigned to each group (EA or non-EA)
Masking Description: all patients undergoing colorectal surgery will be grouped consecutively as epidural anesthesia (EA) or non-EA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA group (Other): patients with colorectal surgery that willl be performed epidural anesthesia
  Interventions: Procedure: epidural anesthesia
- non -EA group (No Intervention): patients with colorectal surgery that willl be performed only general anesthesia

INTERVENTIONS:
Procedure: epidural anesthesia — epidural anesthesia through epidural injection of a local anaesthetic combined with an opioid
  Arms: EA group

SUMMARY:
The use of epidural analgesia (EA) has been suggested as an integral part of an enhanced recovery program for colorectal surgery. However, the effects of EA on postoperative ileus remain controversial. Some authors suggest that EA has beneficial effects for postoperative outcome and hospital stay, whereas others have reported that the role of EA in the modern perioperative care of patients undergoing open colorectal surgery has been limited. Therefore, the investigators aimed to investigate the effect of EA on postoperative outcome, particularly postoperative ileus and hospital stay in patients with colorectal surgery.

DETAILED DESCRIPTION:
In 2016, results of Cochrane review of 22 trials on the efficacy of EA in patients undergoing abdominal surgery showed that an epidural containing a local anesthetic, with or without the addition of an opioid, accelerated the return of gastrointestinal transit (high quality of evidence) and no difference in the incidence of vomiting or anastomotic leak (low quality of evidence). For open surgery, an epidural containing a local anaesthetic would reduce the length of hospital stay (very low quality of evidence).

However, in a recent analysis from American College of Surgeons revealed that the use of EA did not improve postoperative recovery after elective colectomy in their analysis and was associated with increased postoperative ileus and prolonged hospital stay after open colectomy.

In this study, the investigators aimed to compare the efficacy of EA to reduce the postoperative ileus and hospital stay, as well in the patients undergoing colorectal surgery. This prospective randomized study planned to include 100 consecutive patients with colorectal disorders.

ELIGIBILITY:
Inclusion Criteria:

* undergoing colorectal surgery due to both benign and malign disorders
* no contraindication for epidural anesthesia

Exclusion Criteria:

* drug use (psychotropic drugs etc) that may cause paralytic ileus
* immobile patients that ERAS protocol can not be applied on
* Anticoagulated patients with the risk of epidural hematoma,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
postoperative ileus | up to 4 days
  obstipation and intolerance of oral intake due to nonmechanical factors that disrupt propulsive activity of the gastrointestinal system following colorectal surgery..Obstipation was defined as abdominal distention or/and pain at physical examination and difficulty passing gas postoperatively. Intolerance of oral intake was defined as nause or vomiting associated with food intake
prolonged postoperative ileus | up to 10 days
  inability to tolerate oral intake, two or more of nause/ vomiting requiring cessation of oral diet or/and nasogastric decompression and intravenous support, and absence of flatus prolonging hospitalization beyond discharge goal..Prolonged PO was defined as by the postoperative day 5, in case of persistent symptoms mentioned above and radiological confirmation of ileus on plain abdominal film showing multiple distended loops with air and/or fluid and air in both small intestines and large intestines.

SECONDARY OUTCOMES:
hospital stay | up to 1 year
  time from the day of surgery to day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: pinar yazici, Principal Investigator — sisli etfal training and research hospital
Locations (1):
- Pinar Yazici, Istanbul, Other, Turkey (Türkiye)